CLINICAL TRIAL: NCT01755988
Title: Effectiveness of an Interactive Web-based Platform and a Disease Specific Information Website in Patients With Heart Failure: a 3-arm Randomised Trial.
Brief Title: Effectiveness of a Website and Telemonitoring in Patients With Heart Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Foundation: Zorg Binnen Bereik (Unknown)
Responsible Party: Principal Investigator, F.H. Rutten, Dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-456
Record Dates: First submitted 2012-12-12; First posted 2012-12-24 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure
Keywords: Telemedicine; Heart Failure; Self care; Quality of life; Mortality; Hospitalization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (No Intervention)
- Educational website. (Experimental): Educational website (in addition to usual care).
  Interventions: Other: Educational website (in addition to usual care).
- Website and interactive platform with telemonitoring. (Experimental): Adjusted care pathway, including both the educational website and an interactive web-based platform with telemonitoring facilities. In this arm all routine consultations with heart failure nurses and general practitioner will be substituted by this combination of telemonitoring facilities connected to an interactive web-based platform plus the Dutch version of the European Society of Cardiology (ESC) website on heart failure.
  Interventions: Other: Website and interactive platform with telemonitoring.

INTERVENTIONS:
Other: Educational website (in addition to usual care).
  Arms: Educational website.
Other: Website and interactive platform with telemonitoring.
  Arms: Website and interactive platform with telemonitoring.

SUMMARY:
The number of people with heart failure is increasing in the western world. Mainly due to better treatment of myocardial infarctions and ageing of the population. The amount of health care workers is unfortunately not increasing. We want to investigate how two electronic devices (a website and an interactive web-based platform) influence the self-care, quality of life, hospitalizations and mortality by delivering care from a distance. We also want to investigate if a higher quality of care is delivered despite of less frequent visits to a nurse and/or doctor. The study takes place in the Netherlands and is a randomized trial. Patients with heart failure, registered by an outpatient heart failure clinic or general practitioner can take part. They will be randomized to 3 groups: group 1 receives standard care, group 2 receives standard care with the website, group 3 receives an adjusted care pathway, with both the website and the interactive web-based platform connected to a telemonitoring system. In this group all routine consultations with heart failure nurses and general practitioner will be substituted by this device.

ELIGIBILITY:
Inclusion Criteria:

* heart failure established according to the guidelines of the European Society of Cardiology, and confirmed with echocardiography at least three months earlier. The three month period is used to allow for enough time for essential education and initiation of treatment.
* Sufficient cognitive and physical function to understand the aim of the study and perform or undergo the required measurements and sign informed consent.
* Aged 18 years or over.

Exclusion Criteria:

* Non-availability of internet and e-mail.
* Inability to work with internet and e-mail.
* Inability of the patient and his/her family or care takers to read and understand Dutch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in self-care behaviour measured with the validated European Heart Failure Self Care Behaviour Scale(EHFScB scale) | at 3, 6 and 12 months
  The EHFScB measures the behaviour heart failure patients undertake to maintain life, healthy functioning, and well-being. This includes behaviours like adherence to medication, diet and exercise, as well as self-management of symptoms, but it also refers to behaviours such as daily weighing to assess fluid retention and seeking assistance when symptoms occur. The EHFScB is a nine items presented on a 5 point scale.
Change in health related quality of life measured with the generic short-form health survey with 36 questions (SF36), EuroQol five Dimensions (EQ-5D) and the disease-specific Minnesota Living with Heart Failure Questionnaire (MLHFQ) | at 3, 6 and 12 months
  The SF36 is composed of 36 questions with standardized response options, organized in eight multi-item scales: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems and general mental health.
  EQ-5D is a generic questionnaire of health for clinical and economic appraisal and consists of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). Each dimension has 5 levels: from no problems, to severe problems. The MLHFQ is a validated questionnaire and consists of 21 items on patient perceptions concerning the effects of congestive heart failure on their physical, psychologic and socioeconomic lives. Response options are presented as 6 point scale.

SECONDARY OUTCOMES:
Number of patients who died of all causes | at 12 months
Number of heart failure related hospitalisations | at 12 months
Duration of heart failure related hospitalisations | at 12 months
Change in disease specific knowledge measured with the Dutch Heart Failure knowledge scale. | 3, 6 and 12 months
  The Dutch Heart Failure knowledge scale is a 15 item scale that covers items concerning heart failure knowledge in general, knowledge of heart failure treatment (including diet and fluid restriction) and heart failure symptoms and symptom recognition.
Change in heart function measured with blood values. | 6 and 12 months
  N-terminal pro B-type natriuretic peptide (NT-proBNP) levels, renal function ('estimated Glomerular Filtration Rate '(eGFR)) will be used to determine the heart function.
Change in use of website. | 3, 6 and 12 months
  The 'use of website' containing 4 questions targeting how often and how long patients are visiting the website and which parts specifically.
Cost-effectiveness | at 12 months
  To help calculate the cost-effectiveness of the interventions, use of medication, health care use (e.g. hospitalisations, visits to the general practitioner, the outpatient clinics, emergency department and admission to nursing homes) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Arno W Hoes, Dr. MD, Study Director — University Medical Center Utrecht (UMC Utrecht); Frans H Rutten, Dr. MD, Principal Investigator — University Medical Center Utrecht (UMC Utrecht)
Locations (4):
- Netherlands (4):
  - Amstelland hospital, Amstelveen
  - Rijnstate hospital, Arnhem
  - Gelderse Vallei Hospital, Ede
  - Diakonessenhuis hospital, Utrecht

REFERENCES:
- [Derived] Brons M, Ten Klooster I, van Gemert-Pijnen L, Jaarsma T, Asselbergs FW, Oerlemans MIFJ, Koudstaal S, Rutten FH. Patterns in the Use of Heart Failure Telemonitoring: Post Hoc Analysis of the e-Vita Heart Failure Trial. JMIR Cardio. 2023 Jan 31;7:e41248. doi: 10.2196/41248. PMID 36719715
- [Derived] Wagenaar KP, Broekhuizen BDL, Jaarsma T, Kok I, Mosterd A, Willems FF, Linssen GCM, Agema WRP, Anneveldt S, Lucas CMHB, Mannaerts HFJ, Wajon EMCJ, Dickstein K, Cramer MJ, Landman MAJ, Hoes AW, Rutten FH. Effectiveness of the European Society of Cardiology/Heart Failure Association website 'heartfailurematters.org' and an e-health adjusted care pathway in patients with stable heart failure: results of the 'e-Vita HF' randomized controlled trial. Eur J Heart Fail. 2019 Feb;21(2):238-246. doi: 10.1002/ejhf.1354. Epub 2018 Nov 28. PMID 30485612
- [Derived] Wagenaar KP, Broekhuizen BD, Dickstein K, Jaarsma T, Hoes AW, Rutten FH. Effectiveness of an interactive platform, and the ESC/HFA heartfailurematters.org website in patients with heart failure: design of the multicentre randomized e-Vita heart failure trial. Eur J Heart Fail. 2015 Dec;17(12):1310-6. doi: 10.1002/ejhf.413. Epub 2015 Oct 1. PMID 26424105